CLINICAL TRIAL: NCT00822744
Title: An Eight-week, Multicenter, Randomized, Double-blind, Placebo-controlled Dose-finding Study, With Escitalopram (10 mg Daily) as Active Control, to Evaluate the Efficacy, Safety and Tolerability of Three Fixed Doses of SSR411298 (10, 50, or 200 mg Daily) in Elderly Patients With Major Depressive Disorder
Brief Title: An Eight-week Study of SSR411298 as Treatment for Major Depressive Disorder in Elderly Patients
Acronym: FIDELIO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DFI10560; 2008-001718-26 (EudraCT Number)
Record Dates: First submitted 2009-01-13; First posted 2009-01-14 (Estimated); Last update posted 2013-03-15 (Estimated); Status verified 2013-03

CONDITIONS: Major Depressive Disorder
Keywords: Depression; Major Depressive Episode; Antidepressant
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Escitalopram

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- SSR411298 10 mg (Experimental): SSR411298 10 mg, one capsule once daily for 8 weeks
  Interventions: Drug: SSR411298
- SSR411298 50 mg (Experimental): SSR411298 50 mg, one capsule once daily for 8 weeks
  Interventions: Drug: SSR411298
- SSR411298 200 mg (Experimental): SSR411298 200 mg, one capsule once daily for 8 weeks
  Interventions: Drug: SSR411298
- Escitalopram 10 mg (Active Comparator): Escitalopram 10 mg, one capsule once daily for 8 weeks
  Interventions: Drug: Escitalopram
- Placebo (Placebo Comparator): Placebo (for SSR411298), one capsule once daily for 8 weeks
  Interventions: Drug: Placebo (for SSR411298)

INTERVENTIONS:
Drug: SSR411298 — Form: capsule
  Route: oral administration with food
  Arms: SSR411298 10 mg; SSR411298 200 mg; SSR411298 50 mg
Drug: Escitalopram — Form: capsule (commercial escitalopram tablets were encapsulated within opaque capsules)
  Route: oral administration with food
  Arms: Escitalopram 10 mg
Drug: Placebo (for SSR411298) — Form: capsule
  Route: oral administration with food
  Arms: Placebo

SUMMARY:
The primary objective of this study is to evaluate the efficacy of 3 fixed doses of SSR411298 (10, 50 or 200 mg daily) compared to placebo, in elderly patients with Major Depressive Disorder (MDD), based on the 17-item Hamilton Depression Rating Scale.

Secondary objectives are:

* To evaluate the tolerability and safety of an 8-week treatment with SSR411298 versus placebo in elderly patients with MDD.
* To evaluate the effect of SSR411298 on disability, anxiety, cognitive function, sleep, pain and somatic symptoms related to depression, and bone markers.
* To assess SSR411298 plasma concentrations.
* To assess plasma endocannabinoid concentrations.

DETAILED DESCRIPTION:
The study period for a participants is approximately 10 weeks including a screening up to 1 week, 8-week treatment and 1-week follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Elderly patient with recurrent Major Depressive Disorder

Exclusion Criteria:

* Duration of current depressive episode greater than 2 years;
* Mild depression as measured by standard clinical research scales;
* Cognitive disturbance;
* Significant suicide risk;
* Other psychiatric conditions that would obscure the results of the study;
* History of failure to respond to antidepressant treatment.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 527 (Actual)
Dates: Start 2008-12; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
17-item Hamilton Depression Rating Scale (HAM-D) total score | 8 weeks (from D-1 (before randomization) up to D56)
  The HAM-D consists of 17 items assessing signs and symptoms of depression. All items are scored with a severity rating from 0 (not present) to 2 or 4 (very severe), depending on the item. The minimum and maximum possible scores are 0 and 52, respectively.

SECONDARY OUTCOMES:
Montgomery-Asberg Depression Rating Scale (MADRS) total score | 8 weeks (from D-1 (before randomization) up to D56)
  The MADRS consists of 10 items assessing signs and symptoms of depression. All items are scored with a severity rating from 0 (not present) to 6 (most severe). The minimum and maximum possible scores are 0 and 60, respectively.
Clinical Global Impression (CGI) scores | D-1 (before randomization) and D56
  The CGI-1 Severity of Illness score is rated on a 1 to 7 point scale.
  The CGI-2 Improvement score is a component of the CGI; the Improvement score captures the investigator's clinical impression regarding global improvement (or worsening) on a 7-point scale.
HAM-D depressed mood item score, factor scores and core item score | 8 weeks (from D-1 (before randomization) up to D56)
Geriatric Depression Scale (GDS) total score | D-1 (before randomization) and D56
  The GDS is a 15-item self report scale used to assess the more specific aspects of depression in elderly depressed patients.
Sheehan Disability Scale (SDS) total score | D-1 (before randomization) and D56
  The SDS contains 3 questions, which assesses interference in three domains, work and school, family life and home responsibilities, and social life. Each question is answered on a 10-point Likert Scale.
Hamilton Anxiety Rating scale (HAM-A) total score | D-1 (before randomization) and D56
  The HAM-A consists of 14 items assessing signs and symptoms of anxiety. All items are scored with a severity rating from 0 (not present) to 2 or 4 (very severe), depending on the item. The minimum and maximum possible scores are 0 and 56 respectively.
Overview of Adverse Events (AE) | up to 9 weeks (from first study drug intake up to 7 days after last study drug intake)
SSR411298 plasma concentration | predose and 3-5 hours after study drug intake on Day 21 and Day 56
  Plasma concentrations of SSR411298 are determined by a validated liquid chromatography tandem mass spectrometry method with a lower limit of quantification of 10 ng/mL.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (7):
- Sanofi-Aventis Administrative Office, Santiago, Chile
- Sanofi-Aventis Administrative Office, México, Mexico
- Sanofi-Aventis Administrative Office, Bucharest, Romania
- Sanofi-Aventis Administrative Office, Moscow, Russia
- Sanofi-Aventis Administrative Office, Brastislava, Slovakia
- Sanofi-Aventis Administrative Office, Midrand, South Africa
- Sanofi-Aventis Administrative Office, Kiev, Ukraine